CLINICAL TRIAL: NCT01262378
Title: Clinical Outcome of the Seroma Amount Using the Harmonic vs the HF Knife for Surgery According to Lockwood and Abdominoplastic Surgery: A Prospective Controlled Study
Brief Title: Harmonic vs HF Knife in Patients Requiring Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asklepios proresearch (Industry)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Dr. Klaus Mueller, Asklepios Klinik Wandsbek
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASK # 1557; 2909 (Other: Ethics committee der Aerztekammer Hamburg)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2010-12

CONDITIONS: ABDOMINAL SUBCUTANEOUS FAT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Harmonic knife (Other): surgery using the Harmonic knife
  Interventions: Procedure: abdominal plastic surgery
- HF knife (Active Comparator)
  Interventions: Procedure: abdominal plastic surgery

INTERVENTIONS:
Procedure: abdominal plastic surgery — Surgery for ABDOMINAL SUBCUTANEOUS FAT

SUMMARY:
Prospective, non-randomized, controlled study to investigate the clinical outcome of surgery using the Harmonic knife vs the HF knife in patients requiring abdominoplastic surgery or body lift (Lockwood)

DETAILED DESCRIPTION:
Aim of the study is to measure amount of seroma in each interventional arm.

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* willing to give consent
* indication for abdominoplastic surgery
* no contraindication for general anaesthesia

Exclusion Criteria:

* Smoking more than 10 p/day
* Diabetes mellitus I or II
* known neoplasms
* not willing or able to conform with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
amount of seroma | first post operative day until hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Asklepios Klinik Wandsbek, Hamburg, Germany